CLINICAL TRIAL: NCT00152152
Title: Use of Radiostereometric Analysis (RSA) for Measuring Spinal Motion Following Lumbar Spinal Surgery
Brief Title: Use of Radiostereometric Analysis Beads (RSA) to Measure Motion in the Spine, Following Lumbar Spinal Surgery
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: DePuy-Acromed, Inc. (Industry)
Other Study IDs: SUNY UMU IRB# 4715
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Spinal Fusion; Lumbar Discectomy
Keywords: spinal motion; tantalum beads

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Radiostereometric Analysis beads inserted during surgery

SUMMARY:
Radiostereometric Analysis (RSA) is a new imaging technique used to measure motions in the spine. It provides more accurate measurements that could help in diagnosing problems in the spine earlier than standard xray techniques.

DETAILED DESCRIPTION:
Assessment of segmental spinal motion has been and continues to be a difficult clinical problem. X-ray measurement error of up to 10 degrees for simple measurements for flexion, extension and side bending have been recorded. It is extremely difficult to measure small changes in vertebral alignment that may prove to have clinical significance. The measurement accuracy of the RSA technique far exceeds any manual techniques to date. RSA allows the surgeon to monitor spatial relationships within the spine over time with a much higher accuracy then conventional techniques.

This is a non-randomized prospective study design looking at the use of RSA in spinal surgery patients. Subjects in this study will undergo their indicated surgery. Prior to closure, they will be implanted with tantalum beads, which will serve as landmarks when the RSA film pairs are taken post-operatively. The subjects will have standard post-operative x-rays 6 weeks-3 months post-op and again at 12 months post-op. Yearly visits after this are anticipated for 5-10 years with proper funding.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Spinal fusion or discectomy

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2002-10; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E. Fredrickson, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States